CLINICAL TRIAL: NCT03437187
Title: The Beneficial Effect of Quadratus Lumborum Block After Laparoscopic Cholecystectomy in Day-Case Surgery: A Randomized Controlled Trial
Brief Title: The Beneficial Effect of Quadratus Lumborum Block After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Responsible Party: Principal Investigator, Jan Sverre Vamnes, Senior consultant, MD, Ph.D., Ostfold Hospital Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1812
Record Dates: First submitted 2018-01-22; First posted 2018-02-19 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Cholecystectomy; Quadratus Lumborum Block
MeSH Terms: interventions — Cholecystectomy; Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Masking Description: Information connecting the patients to the data are kept locked and will be destroyed after the end of the investigation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cholecystectomy without nerve blocks (Other): Cholecystectomy, enteral and parenteral analgesics
  Interventions: Procedure: Cholecystectomy
- Cholecystectomy with placebo nerve block (Placebo Comparator): Cholecystectomy, NaCl as a placebo Quadratus lumborum block
  Interventions: Procedure: Cholecystectomy
- Cholecystectomy with naropin nerve block (Active Comparator): Cholecystectomy, Quadratus lumborum block with naropin
  Interventions: Procedure: Cholecystectomy

INTERVENTIONS:
Procedure: Cholecystectomy — Laparoscopic technique
  Other Names: Quadratus lumborum block with Naropin; Quadratus lumborum block with Nacl; Traditional analgesics

SUMMARY:
The enhanced recovery after surgery and laparoscopic approach is essential after day-case surgery. The patients want to go home early without pain and nausea, and the hospitals need the post-operative capacity for more patients. Many patients have pains, nausea and vomiting postoperatively. Postoperative pain is an expected but undesirable effect after an operation. The aim of the study is to find out if a bilateral quadratus lumborum block has a beneficial effect after a cholecystectomy.

DETAILED DESCRIPTION:
QLB (quadratus lumborum block) is a recommended multimodal method of reducing postoperative pain in laparoscopic and open surgery. Quadratus lumborum block for postoperative pain after caesarean section 2015). Transversus abdominis plane (TAP) block seems to be feasible and effective in postoperative pain control without increasing morbidity in cholecystectomy. QLB is also performed as one of the perioperative pain management procedures in abdominal surgery. It is regarded as an effective analgesic tool The dermatomal effects of QLB reach higher than the TAP block and might explain the better effect of the QLB than TAP blocks on postoperative pain after caesarean delivery. A randomized double blinded clinical trial with TAP block in patients scheduled for cholecystectomy is performed, but there is no good data for the QLB. For this study the investigators standardize the type of surgery to be laparoscopic day-case cholecystectomy, and we use the anterior (transmuscular) QLB.

Power and Sample Size Calculator The number of patients required for the study was calculated on the basis of opioid consumption. The investigators are interested in a reduction by 20% in the group given QLB. Assuming α=0,05, the calculation shows a need of 69 patients (23 in each group) to achieve a power of 80% (β=0.2).

75 adult patients scheduled for cholecystectomy have to be included. Subcutaneous wound infiltration at the end of surgery in all patients with ropivacaine 2 mg/ml, 10 ml. Maximum allowed dosis is 3 mg/kg BW (BodyWeight). Dosis reduction if BW<70 kg. All three groups receive necessary analgesics oral or parenteral.

Premedication: Paracetamol 2g and Diklofenak 100 mg

General anesthesia: TCI (Target Control of Infusion): Propofol and Remifentanil, Ondansetron 4 mg and Decadron 8 mg iv preoperatively. Oxycodon 5 mg iv at the end of the procedure.

Surgical procedure: Cholecystectomy, laparoscopic and day-case.

Postoperatively:

* Oral paracetamol and codeine-fixed combination up to 1000 mg and 60 mg, respectively, every 6 h
* In case of insufficient analgesia, as judged by the patient, oxycodon 1 - 5 mg IV.
* When nausea and vomiting occur postoperatively, ondansetron 4 mg IV administers as the drug of first choice followed by droperidol 0,625 mg IV if the nausea/vomiting persists.

Collected data:

* Postoperative pain at rest and during activity evaluates by a 0 - 10 scale (NRS) on admission to recovery, and every hour until discharge.
* Rescue analgesic consumption during 0 to 4, 4 to 24 and 24 to 48 h.
* Nausea and vomiting record by the same 0 - 3 scale (none, slight, moderate, strong) during recovery
* Time of postoperative mobilization with corresponding pain score.
* Time of discharge-to-home readiness according to standard criteria, including stable vital signs, no bleeding from the surgical site, ability to void, absence of excessive nausea and pain, and ability to dress and walk without support.
* Side effects including nausea and/or vomiting (0 to 4, 4 to 24, and 24 to 48 h), and other side effects and symptoms of LA (Local Anaesthetic) toxicity.

Telephone interview at 24 h and 48 h

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 Years
* BMI 20-35
* ASA physical status I-II

Exclusion Criteria:

* Allergy to local anaesthetics
* Chronic pain requiring opioid analgesics
* Patients with atrioventricular block II
* Patients treated with class III antiarrhythmics
* Patients with severe renal and/or hepatic disease
* A coagulation disorder
* An infection at the LA injection place

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
Use of analgesics -"change" is being assessed | 1 week (0-4hrs) (4-24hrs) (24-48hrs)
  Amount of analgesics used postoperative

SECONDARY OUTCOMES:
Pain at the incision site - "change" is being assessed | 48 hours (0-4hrs) (4-24hrs) (24-48hrs)
  NRS (Numeric Rating Scale; 0 - 10) 0 = no pain, 10 = severe pain
Deep pain and pain on coughing - "change" is being assessed | 48 hours (0-4hrs) (4-24hrs) (24-48hrs)
  NRS (Numeric Rating Scale; 0 - 10) 0 = no pain, 10 = severe pain
Nonsteroidal anti-inflammatory drug consumption - "change" is being assessed | 48 hours(0-4hrs) (4-24hrs) (24-48hrs)
  Amount of different medicaments in mg
Postoperative nausea and vomiting - "change" is being assessed | 48 hours(0-4hrs) (4-24hrs) (24-48hrs)
  0-3 score where 0=none, 1=little nausea, 2=can not eat, 3=vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Ostfold Hospital Trust, Moss, Grålum, Østfold fylke, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Borglum J, Gogenur I, Bendtsen TF. Abdominal wall blocks in adults. Curr Opin Anaesthesiol. 2016 Oct;29(5):638-43. doi: 10.1097/ACO.0000000000000378. PMID 27429253
- [Result] Blanco R, Ansari T, Riad W, Shetty N. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block for Postoperative Pain After Cesarean Delivery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):757-762. doi: 10.1097/AAP.0000000000000495. PMID 27755488
- [Result] El-Dawlatly AA, Turkistani A, Kettner SC, Machata AM, Delvi MB, Thallaj A, Kapral S, Marhofer P. Ultrasound-guided transversus abdominis plane block: description of a new technique and comparison with conventional systemic analgesia during laparoscopic cholecystectomy. Br J Anaesth. 2009 Jun;102(6):763-7. doi: 10.1093/bja/aep067. Epub 2009 Apr 17. PMID 19376789
- [Result] Murouchi T, Iwasaki S, Yamakage M. Quadratus Lumborum Block: Analgesic Effects and Chronological Ropivacaine Concentrations After Laparoscopic Surgery. Reg Anesth Pain Med. 2016 Mar-Apr;41(2):146-50. doi: 10.1097/AAP.0000000000000349. PMID 26735154
- [Result] Petersen PL, Stjernholm P, Kristiansen VB, Torup H, Hansen EG, Mitchell AU, Moeller A, Rosenberg J, Dahl JB, Mathiesen O. The beneficial effect of transversus abdominis plane block after laparoscopic cholecystectomy in day-case surgery: a randomized clinical trial. Anesth Analg. 2012 Sep;115(3):527-33. doi: 10.1213/ANE.0b013e318261f16e. Epub 2012 Jul 4. PMID 22763903
- [Result] Ueshima H, Otake H, Lin JA. Ultrasound-Guided Quadratus Lumborum Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:2752876. doi: 10.1155/2017/2752876. Epub 2017 Jan 3. PMID 28154824